CLINICAL TRIAL: NCT05009264
Title: Treating Trigger Points: Comparing Muscle Energy Technique vs. Lidocaine Needling Technique for Pain Control and Quality of Life Measurements
Brief Title: OMTrigger Inject- Treating Trigger Points: Comparing Muscle Energy Technique vs. Lidocaine Needling Technique
Status: Terminated | Type: Observational
Why Stopped: Principal investigator no longer working at our facility
Sponsor: AtlantiCare Regional Medical Center (Other)
Collaborators: Philadelphia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 2021-1045
Record Dates: First submitted 2021-07-16; First posted 2021-08-17 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Tocopherols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OMT Group: This group will receive OMT muscle energy as treatment for myofascial pain syndrome
  Interventions: Procedure: OMT
- Injection Group: This group will receive lidocaine injections for myofascial pain syndrome
  Interventions: Procedure: OMT

INTERVENTIONS:
Procedure: OMT — OMT will be performed on identified areas of trapezius trigger points
  Other Names: muscle energy

SUMMARY:
The primary aim of this study is to determine if osteopathic manipulative treatment is as effective to traditional lidocaine injection technique in treating myofascial trigger points in regard to post intervention pain intensity and quality of life.

DETAILED DESCRIPTION:
Myofascial pain syndrome is one of the most common musculoskeletal disorders seen in the aging US population. Its characterized by myofascial trigger points (MTPs) which were defined as hyperirritable nodules in a taut band of skeletal muscle, associated with pain on manual stretching, contraction, or stimulation of the muscle. Trigger points are further classified into active and latent based on their clinical features. Active MTPs are characterized by spontaneous pain at rest with referred pain on palpation whereas latent MTPs produce pain on palpation in addition to restriction of range of motion.

Currently, there are a variety of treatment options for MTPs including lidocaine injections, dry needling, osteopathic manipulative treatment, massage therapy, ultrasound therapy etc. There has been a lot of research investigating the safety and efficacy of dry needling and lidocaine trigger point injection techniques in treating MTPs. It was found that dry needling and lidocaine injections were both equally effective in reducing symptoms associated with MTPs as it was the mechanical disruption of the taut fibers due to the needle effect and the depth of adequate penetration that resulted in pain reduction more than the substance actually delivered into the muscle. Some authors also suggested the importance of a local twitch response (LTR); which is an observable contraction of the taut part of muscle band upon stimulation, during dry needling technique as being pertinent for maximum effectiveness. However, a recent systemic review found that LTR during dry needling treatment was unnecessary and not required for management of myofascial pain syndrome.

On the other hand, there has been fewer research investigating the effects of manual treatment on trigger points. Reasearchers had initially treated trigger points with ischemic compression but later changed their recommendation to applying gentle digital pressure to trigger points. A recent study done on traction-compression-stretch technique (TTCE) compared with ischemic compression showed some, albeit minor, increased outcome measures (pain pressure threshold) warranting clinical investigation. Another study compared active release and muscle energy techniques in treating latent trigger points of the upper trapezius and found that both techniques were equally effective in increasing cervical range of motion and decreasing pain and upper trapezius thickness. Other studies have also shown interest in similar osteopathic manipulative techniques such as counterstrain, myofascial release, facilitated positional release and high velocity-low amplitude thrust techniques in treating trigger points.

Studies have showed that the upper trapezius is one of the most common muscles affected by myofascial pain syndrome leading to referred pain manifesting as headaches and stiff neck.

Currently, there is no consensus as to which treatment method is superior, with the decision to treat in a certain way largely based upon the training received by the individual physician rather than the characteristics of the trigger point itself. There are no studies to date evaluating the efficacy of the various treatment options specifically osteopathic manipulative treatment vs. trigger point injections. Thus, the intention of the present study is to determine the efficacy rates of muscle energy techniques vs. lidocaine injections in treating MTPs in the upper trapezius region.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will only be recruited into the study if participants have met all the following criteria:

  * Ages between 25 and 75 years.
  * Previous or current diagnosis of MTrP in the upper trapezius region according to the criteria in reference
  * 1 active/latent MTrP in the upper trapezius region

The diagnostic criteria to establish myofascial trigger point is adopted from prior investiogators and include:

1. Presence of palpable taut band in the skeletal muscle
2. Presence of hypersensitive tender spot in the taut band
3. Presence of local twitch response upon stimulation of the taut band
4. Reproduction of referred pain upon palpation
5. Presence of spontaneous referred pain pattern

Exclusion Criteria:

* Exclusion criteria: Any subject that exhibits any of the following criteria will excluded from the study:
* Pregnancy or immunocompromise
* Fever/infection
* Previous history of whiplash injury
* Previous history of cervical surgery, cervical radiculopathy, or myelopathy
* Severe disc or cervical lesion
* Evidence of cognitive deficit
* Degenerative or inflammatory disease of the cervical spine or shoulder, fibromyalgia, or neuromuscular diseases
* Use of medications (anticoagulants, anti-inflammatory etc.) or illicit drug use (1 week prior to treatment or follow up)
* Received treatment for MPS a month before the study recruitment

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is a prospective cohort study comprised of participants between ages 25-75 that presented to Atlanticare Regional Medical Center interventional pain department and Philadelphia College of Osteopathic Medicine Osteopathic Clinic between 2021 August and 2021 october with trigger point in the upper trapezius muscle. It is expected that approximately 60 patients will be enrolled to produce approximately 50 evaluable subjects.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Prior to intervention
  0-10, measured using a point system; where 0 = no pain and 10 = maximum pain.
Measurement on quality of life, evaluate neck and upper extremity function. | Prior to intervention
  Utilizing the neck disability index score which is used to evaluate neck and upper extremity function. The total score is divided by number of answered questions, subtracted 1 and multiplied by 25, in a scale score that range from 0 to 100, with higher scale scores indicating more disability.
Pain Intensity | Immediately after intervention
  0-10, measured using a point system; where 0 = no pain and 10 = maximum pain.
Measurement on quality of life, evaluate neck and upper extremity function. | immediately after intervention
  Utilizing the neck disability index score which is used to evaluate neck and upper extremity function. The total score is divided by number of answered questions, subtracted 1 and multiplied by 25, in a scale score that range from 0 to 100, with higher scale scores indicating more disability.
Pain Intensity | 1 week after intervention
  0-10, measured using a point system; where 0 = no pain and 10 = maximum pain.
Measurement on quality of life, evaluate neck and upper extremity function. | 1 week after intervention
  Utilizing the neck disability index score which is used to evaluate neck and upper extremity function. The total score is divided by number of answered questions, subtracted 1 and multiplied by 25, in a scale score that range from 0 to 100, with higher scale scores indicating more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan S Kelly, DO, Principal Investigator — AtlantiCare Regional Medical Center
Locations (1):
- AtlantiCare Regional Medical Center, Atlantic City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a multisite study and information may be shared between the institutions

REFERENCES:
- [Result] Hong CZ, Hsueh TC. Difference in pain relief after trigger point injections in myofascial pain patients with and without fibromyalgia. Arch Phys Med Rehabil. 1996 Nov;77(11):1161-6. doi: 10.1016/s0003-9993(96)90141-0. PMID 8931529

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT05009264/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT05009264/SAP_001.pdf